CLINICAL TRIAL: NCT06035939
Title: Self-Management for Youth Living With Sickle Cell Disease: SMYLS Multi-site Trial
Brief Title: SMYLS Multi-site Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Shannon Phillips, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00127137; 1R01NR020606-01 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Study participants randomized to receive the intervention.
  Interventions: Behavioral: Voice Crisis Alert V2
- Control (Active Comparator): Study participants randomized to receive enhanced usual care (control).
  Interventions: Behavioral: Electronic educational materials

INTERVENTIONS:
Behavioral: Voice Crisis Alert V2 — The mHealth self-management intervention consists of the following components: 1) condition-specific electronic educational materials; 2) pain/symptom monitoring and tracking; 3) health history information documentation; 4) medication tracking; 5) secure messaging with a provider; 6) functioning monitoring and tracking; and 7) transmission of health information (graphs with recorded pain and functioning histories) to a provider.
  Arms: Intervention
Behavioral: Electronic educational materials — The control arm will receive enhanced usual care, which will consist of usual educational materials distributed at the clinic plus a version of the intervention (Voice Crisis Alert V2) that only includes the electronic educational materials.
  Arms: Control

SUMMARY:
The purpose of this study is to find out whether a web-based intervention using a mobile app is helpful for teens and young adults with sickle cell disease (SCD) in learning how to care for and manage their symptoms.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness of and identify barriers and facilitators to the implementation of SMYLS, an mHealth intervention designed to facilitate self-management behaviors in adolescents and young adults (AYA) with sickle cell disease (SCD). Specifically, the investigators propose to determine the effect of the intervention on the primary outcome of self-management behaviors and the secondary outcomes of quality of life, transition readiness, healthcare utilization, and pain interference. In addition, the investigators will explore how patient activation moderates development of self-management behaviors and systemic, structural, and social variables that moderate relationships between patient activation, the primary outcome, and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* documentation in the electronic health record of any type of SCD
* owns mobile device compatible with the intervention
* access to the internet

Exclusion Criteria:

* Plans to relocate outside of study site area in the next 12 months
* Plans to transition to adult care in 12 months or less
* Parent/caregiver or provider report of neurocognitive impairment that precludes ability to use intervention and participate in study
* non-English speaking

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 272 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Self-management behaviors | baseline and 1, 3, 6, 9, 12 months
  Adolescent and young adult self-report using the Transition Readiness Assessment Questionnaire 5th version (TRAQ-5; 20 items). The instrument consists of 5 scales. Individual item scores range from 1 - 5. Scale scores are determined by calculating the average of the item scores within each scale. Higher scores indicate greater transition readiness and self-management behaviors.

SECONDARY OUTCOMES:
Engagement in intervention/control (categorical) | baseline and 1, 3, 6, 9, 12 months
  Categorized into none, low, moderate and high. For intervention arm, categories are based on scope (number of components), duration (number of weeks), and frequency (number of times per week). For control arm, categories are based on duration and frequency as for intervention group parameters.
Engagement in intervention/control (continuous) | Ongoing
  Number of times the application is accessed (intervention = full application; control = educational component only).
Health-related quality of life | baseline and 1, 3, 6, 9, and 12 months
  Adolescent and young adult self report using the Pediatric Quality of Life Inventory (PedsQL) with Sickle Cell Disease Module (43 items). Items are scaled from 0 (Never) to 4 (Almost always). Scores are reverse scored and linearly transformed to a 0 - 100 scale. Higher scores indicate better health-related quality of life.
Number of attended SCD clinic visits | baseline and 1, 3, 6, 9, and 12 months
  Number of attended SCD clinic visits documented in the medical record
Number of ED visits | baseline and 1, 3, 6, 9, and 12 months
  Number of ED visits documented in the medical record
Number of hospitalizations | baseline and 1, 3, 6, 9, and 12 months
  Number of hospitalizations documented in the medical record
Pain interference | baseline and 1, 3, 6, 9, and 12, months
  Adolescent and young adult self report using the Patient Reported Outcomes Measurement Inventory System (PROMIS) Pain Interference v2 Pediatric Short Form (8 items). Raw scores range from 0 - 32 with higher scores indicating greater pain interference.
Transition readiness | baseline and 1, 3, 6, 9, and 12 months
  Adolescent and young adult self report using the Transition Intervention Program - Readiness for Transition (TIP-RFT; 22 items). Scores for each item range from 0 - 4, with a total possible summed score ranging from 0 - 88. Lower scores indicate higher transition readiness.

OTHER OUTCOMES:
Patient activation | baseline and 1, 3, 6, 9, and 12 months
  Moderator variable; adolescent and young adult self-report using the Patient Activation Measure (PAM-13). Raw scores are transformed to a scale of 0 - 100 with 100 being the highest activation level.
Neurocognitive/executive functioning | baseline, 9 months
  Moderator variable; adolescent's parent/caregiver report using the Behavior Rating Inventory of Executive Function, 2nd ed. (BRIEF-2; 12 items). Raw scale scores are transformed to T scores. T scores from 60-64 are mildly elevated problems with executive functioning, T scores from 65-69 are considered potentially clinically elevated problems with executive functioning, and T scores at or above 70 are considered clinically elevated problems with executive functioning.
Social resources and conditions | baseline, 9 months
  Moderator variable; based on residential address using the Child Opportunity Index (COI). 9-month measurement will assess change in address and change in COI. All United States neighborhoods are scored and ranked from lowest to highest opportunity. Five levels of opportunity are used (very low, low, moderate, high, very high) and scores range from 1 (lowest opportunity) to 100 (highest opportunity).
Depressive symptoms | baseline, 9 months
  Moderator variable; adolescent and young adult self report using the Patient Reported Outcomes Measurement Information System (PROMIS) Depressive Symptoms v2 Pediatric Short Form (8 items). Raw scores range from 0 - 32 with higher scores indicating greater depressive symptoms.
Anxiety | baseline, 9 months
  Moderator variable; adolescent and young adult self report using the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety v2 Pediatric Short Form (8 items). Raw scores range from 0 - 32 with higher scores indicating greater anxiety.
Fatigue | baseline, 9 months
  Moderator variable; adolescent and young adult self report using the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue v2 Pediatric Short Form (10 items). Raw scores range from 0 - 40 with higher scores indicating greater fatigue.
Family functioning | baseline, 9 months
  Moderator variable; parent/caregiver of adolescent report using the McMaster Family Functioning Assessment Device (12 items). Items response options range from 1 (strongly agree) to 4 (strongly disagree). All odd items are reverse scored. After reverse scoring, all items are summed. Lower total scores indicate higher levels of family functioning.
Health literacy | baseline, 9 months
  Moderator variable; adolescent and young adult self report using the Newest Vital Sign (NVS; 6 items). Items are scored from 0 - 6 and summed. Total scores of 0 - 1 indicate a high likelihood of limited literacy, 2 - 3 a possibility of limited literacy, and 4 - 6 adequate literacy.
Perceived stigma | baseline, 9 months
  Moderator variable; adolescent and young adult self report using the Child Stigma Scale (8 items). Each item is rated from from 0 (Never) to 4 (Very often). Higher scores indicate greater perceived stigma.
Sleep disturbance | baseline, 9 months
  Moderator variable; adolescent and young adult self report using the Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance v1 Pediatric Short Form (4 items). Raw scores range from 0 - 16 with higher scores indicating greater sleep disturbance.
Perceived discrimination | baseline, 9 months
  Moderator variable; adolescent and young adult self report using the Discrimination subscale of the Interpersonal Processes of Care instrument (2 items). Response options range from 1 (Never) to 5 (Always). Total score is calculated as the mean of responses, with higher scores indicating higher frequency of discrimination.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Phillips S, Martin K, Schlenz AM, Kanter J, Mueller M, Lebensburger J, Galandanci N, Fuh BR, Rivenbark C, Alvarez OA, Hanson RF, Madisetti M, Prentice M, Kelechi TJ. Self-Management for Youth Living with Sickle Cell Disease (SMYLS): A study protocol for a multisite randomized controlled trial testing a behavioral, mHealth app. Contemp Clin Trials. 2025 Nov;158:108103. doi: 10.1016/j.cct.2025.108103. Epub 2025 Oct 4. PMID 41052714